CLINICAL TRIAL: NCT05048810
Title: Clinical Application of 68Ga-DOTA-NT-20.3 in the Early Diagnosis of Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, FengWang, Director of nuclear medicine department, Nanjing First Hospital, Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 68Ga-DOTA-NT-20.3
Record Dates: First submitted 2020-02-06; First posted 2021-09-17 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Pancreatic Ductal Adenocarcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-DOTA-NT-20.3 (Experimental): Subjects will undergo PET imaging using 68Ga-DOTA-NT-20.3.
  Interventions: Radiation: 68Ga-DOTA-NT-20.3

INTERVENTIONS:
Radiation: 68Ga-DOTA-NT-20.3 — In this study, all patients will receive one injection of 68Ga-DOTA-NT-20.3, a PET radiopharmaceutical selective for neurotensin receptor 1 (NTR-1). For the injection, subjects will receive a target dose of 2-4 MBq per kg of body weight as a bolus injection. 68Ga-DOTA-NT-20.3 injection will be followed by a 10 ml saline flush.

SUMMARY:
The purpose of this study is to determine the pharmacokinetics, dosimetry, tolerance, tumor detection rate of 68Ga-DOTA-NT-20.3 in patient with pancreatic ductal adenocarcinoma (PDAC).

DETAILED DESCRIPTION:
This study is design to prospectively investigate the safety and efficacy of 68Ga-DOTA-NT-20.3 in the early diagnosis of pancreatic ductal adenocarcinoma (PDAC). The specific objectives are the determination of pharmacokinetics, dosimetry, tolerance and tumor detection rate of 68Ga-DOTA-NT-20.3 in patient with PDAC. Neurotensin receptor 1 (NTR-1) is the high affinity receptor of Neurotensin (NT), which was found abnormal expression in the early stages of PDAC malignant cell transformation. 68Ga-DOTA-NT-20.3 as a new NTR-1 targeted probe was prepared and showed good uptake on PDAC cell line and animal studies. The study intends to recruit 6 PDAC volunteers to participate in the experiment. Patients were evaluated with 18F-fluorodeoxyglucose (18F-FDG). And then all patients underwent a single-injection with 68Ga-DOTA-NT-20.3, dual-modality imaging protocol consisting of a PET/CT and subsequent PET/MR scan. The follow-up period was followed up to assess safety and effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* patient with pathohistologically proven localized or metastatic PDAC;
* patient aged 18 or older, male or female, who can provide written informed consent for this study;
* patient with complete clinical data.

Exclusion Criteria:

* patient age < 18 years;
* patient with other active cancer;
* patient with PDAC under the treatment blocking NT receptors;
* pregnant or lactating women;
* patient who cannot stay on PET/CT camera for app. 90 minutes;
* patient who cannot stand MRI;
* patient simultaneously participating in another clinical trial;
* patient with HIV, HCV, HVB infection or other serious chronic infection
* patient with serious mental, neurological, cardiovascular, respiratory and other system diseases;
* patient with liver and kidney function (GFR less than 50 ml/min) disease;
* patient with severe severe refractory mental disorder.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-02-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of diagnosis and staging | 3 years
  The presence of non-physiological uptake or uptake in a tissue structure can be considered pathological. The signal intensity of PET indicates the presence and density of NTR-1 in the tissue. The lesion intake is higher than the liver and is classified as clearly positive. The lesion and the surrounding normal tissue ROI, measure the SUV, and calculate the T/B ratio.

SECONDARY OUTCOMES:
NTR-1 receptor expression by histology compared to tracer uptake | 3 years
  Pathological detection of NTR-1 receptor expression in patients' lesions and compared to tracer uptake by PET/CT/MR.
Safety and Tolerability Profile Measured by Adverse Events (AEs) | 3 years
  Safety and tolerability profile for the administration of 68Ga-DOTA-NT-20.3 and positron emission tomography (PET) scanning are measured by number of participants with adverse events (AEs).

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Ph.D, Study Director — Nuclear Medicine Department, Nanjing First Hospital
Locations (1):
- Nanjing First Hospital, Nanjing, China